CLINICAL TRIAL: NCT02731079
Title: Prospective Comparison of Sleeve Gastrectomy Outcomes With Different Stapling Devices
Brief Title: Sleeve Gastrectomy Outcomes With Different Stapling Devices
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study expired before any data was analyzed.
Sponsor: Edna Rath (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Edna Rath, Human Protection Director, William Beaumont Army Medical Center
Organization: William Beaumont Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WB16-08
Record Dates: First submitted 2016-03-30; First posted 2016-04-07 (Estimated); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Morbid Obesity
Keywords: Sleeve gastrectomy stapler Covidien Ethicon bleeding leak
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Covidien (Active Comparator): Group that will have sleeve gastrectomy performed using the Covidien iDrive powered stapler with absorbable polymer membrane staple line reinforcement.
  Interventions: Device: Covidien iDrive
- Ethicon (Active Comparator): Group that will have sleeve gastrectomy performed using the Ethicon Echilon powered stapler with absorbable polymer membrane staple line reinforcement.
  Interventions: Device: Ethicon Echilon

INTERVENTIONS:
Device: Covidien iDrive — Surgery performed with Covidien powered stapler
  Arms: Covidien
Device: Ethicon Echilon — Surgery performed with Ethicon powered stapler
  Arms: Ethicon

SUMMARY:
Sleeve gastrectomy is now the most commonly performed bariatric surgery. While many studies have evaluated factors that may minimize post-operative hemorrhage and staple-line leak, the investigators are unaware of any studies that compare outcomes between devices from the two main stapler manufacturers used in this surgery, Covidien and Ethicon. The purpose of this study is to compare intraoperative characteristics, such as time to create sleeve, intraoperative bleeding, and time needed to load each cartridge, and post-operative characteristics, such as any complication requiring readmission (leak or hemorrhage), further surgical intervention, and weight loss, between patients who underwent sleeve gastrectomy with Covidien devices and Ethicon devices. Currently the investigators predominantly use whatever device is cheaper, but cost should not be the primary decisive factor if one device is superior to the other. If one device has better clinical outcomes, it should be the preferred device regardless of cost. If neither proves superiority, the investigators can justify using cost to determine which device to use in patient care.

DETAILED DESCRIPTION:
New bariatric patients who have elected for a sleeve gastrectomy as part of standard of care will be invited to participate in the study during the bariatric clinic at William Beaumont Army Medical Center. Patients who meet the inclusion criteria will be invited to participate in the study. These patients will be consented in the bariatric clinic by a research coordinator (Doreen Bandari-Spaulding) or physician listed on the study if the coordinator is unavailable.

Three folders will be made, one for each bariatric surgeon, and 25 Covidien cards and 25 Ethicon cards will be placed into each for a total of 150 patients. All bariatric surgeons are trained and familiar with both devices. Once consented, a card will be removed at random to determine which stapler will be used. Bioabsorbable staple line reinforcement will be utilized with both staplers. Once in the operating room, the case start time, time from first staple firing to completion of sleeve, total stapler loads required, number of staple misfires, character of any staple line bleeding, and time for tech to load each cartridge will be recorded on a data collection sheet by a research resident, listed as an associative investigator on this protocol. The subject's post-operative course will follow the bariatric protocol. During follow-up, they will be monitored for weight loss, post-operative complications, and any other required interventions. This information will be obtained by reviewing the subject's medical record after follow-up appointments. Per the institutional bariatric protocol, subjects will follow-up at 3 weeks, 6 weeks, 3 months, 6 months, and annually. If a subject withdraws consent for the study prior to surgery, they will still receive surgery and perioperative treatment in line with institutional protocol, and they will be withdrawn and create a vacancy for a new subject. If a subject withdraws consent after surgery, data collection will cease for that subject. The investigators will clarify whether they want all data to be removed from the study or if they simply want no more data to be entered into the study and abide by their wishes, and they will remain in the original randomized group in accordance with intention-to-treat principles.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained and signed from each subject
2. Age ≥ 18 years
3. Requirement for agreement to avoid conception
4. BMI >40
5. BMI >35 with obesity-related co-morbidity
6. Pre-operative psychiatric evaluation
7. Pre-operative laboratory studies that fail to demonstrate secondary cause of obesity
8. Full course of triple therapy for patients with Helicobacter pylori on upper endoscopy

Exclusion Criteria:

1. Pregnancy- Patients are not eligible for bariatric surgery, and if they become pregnant after surgery, they would present confounding variables and alter weight loss
2. Tobacco use within one month of surgery or any time within study period- Most staff will not perform bariatric surgery on active smokers as it negatively impacts healing
3. Prior bariatric surgery- Makes repeat bariatric surgery more difficult and could increase risk of complications
4. Inflammatory bowel disease- Rare diagnosis that may increase chance of complications, thus confounding results
5. Active duty military- Not eligible for bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric P Ahnfeldt, DO, Principal Investigator — Residency Program Director
Locations (1):
- William Beaumont Army Medical Center, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] Nguyen NT, Nguyen B, Gebhart A, Hohmann S. Changes in the makeup of bariatric surgery: a national increase in use of laparoscopic sleeve gastrectomy. J Am Coll Surg. 2013 Feb;216(2):252-7. doi: 10.1016/j.jamcollsurg.2012.10.003. Epub 2012 Nov 21. PMID 23177371
- [Background] Marceau P, Hould FS, Simard S, Lebel S, Bourque RA, Potvin M, Biron S. Biliopancreatic diversion with duodenal switch. World J Surg. 1998 Sep;22(9):947-54. doi: 10.1007/s002689900498. PMID 9717420
- [Background] Ren CJ, Patterson E, Gagner M. Early results of laparoscopic biliopancreatic diversion with duodenal switch: a case series of 40 consecutive patients. Obes Surg. 2000 Dec;10(6):514-23; discussion 524. doi: 10.1381/096089200321593715. PMID 11175958
- [Background] Regan JP, Inabnet WB, Gagner M, Pomp A. Early experience with two-stage laparoscopic Roux-en-Y gastric bypass as an alternative in the super-super obese patient. Obes Surg. 2003 Dec;13(6):861-4. doi: 10.1381/096089203322618669. PMID 14738671
- [Background] ASMBS Clinical Issues Committee. Updated position statement on sleeve gastrectomy as a bariatric procedure. Surg Obes Relat Dis. 2012 May-Jun;8(3):e21-6. doi: 10.1016/j.soard.2012.02.001. Epub 2012 Feb 10. No abstract available. PMID 22417852
- [Background] D'Ugo S, Gentileschi P, Benavoli D, Cerci M, Gaspari A, Berta RD, Moretto C, Bellini R, Basso N, Casella G, Soricelli E, Cutolo P, Formisano G, Angrisani L, Anselmino M. Comparative use of different techniques for leak and bleeding prevention during laparoscopic sleeve gastrectomy: a multicenter study. Surg Obes Relat Dis. 2014 May-Jun;10(3):450-4. doi: 10.1016/j.soard.2013.10.018. Epub 2013 Nov 12. PMID 24448100
- [Background] Gentileschi P, Camperchioli I, D'Ugo S, Benavoli D, Gaspari AL. Staple-line reinforcement during laparoscopic sleeve gastrectomy using three different techniques: a randomized trial. Surg Endosc. 2012 Sep;26(9):2623-9. doi: 10.1007/s00464-012-2243-2. Epub 2012 Mar 23. PMID 22441975
- [Background] Glaysher M, Khan OA, Mabvuure NT, Wan A, Reddy M, Vasilikostas G. Staple line reinforcement during laparoscopic sleeve gastrectomy: does it affect clinical outcomes? Int J Surg. 2013;11(4):286-9. doi: 10.1016/j.ijsu.2013.02.015. Epub 2013 Feb 28. PMID 23459188
- [Background] Sroka G, Milevski D, Shteinberg D, Mady H, Matter I. Minimizing Hemorrhagic Complications in Laparoscopic Sleeve Gastrectomy--a Randomized Controlled Trial. Obes Surg. 2015 Sep;25(9):1577-83. doi: 10.1007/s11695-015-1580-3. PMID 25596939
- [Background] Gagner M, Buchwald JN. Comparison of laparoscopic sleeve gastrectomy leak rates in four staple-line reinforcement options: a systematic review. Surg Obes Relat Dis. 2014 Jul-Aug;10(4):713-23. doi: 10.1016/j.soard.2014.01.016. Epub 2014 Jan 28. PMID 24745978
- [Background] Huang R, Gagner M. A Thickness Calibration Device Is Needed to Determine Staple Height and Avoid Leaks in Laparoscopic Sleeve Gastrectomy. Obes Surg. 2015 Dec;25(12):2360-7. doi: 10.1007/s11695-015-1705-8. PMID 26024735

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in the US scheduled to have a sleeve gastrectomy.
Groups:
- Covidien: Group that will have sleeve gastrectomy performed using the Covidien iDrive powered stapler with absorbable polymer membrane staple line reinforcement. Covidien iDrive: Surgery performed with Covidien powered stapler
- Ethicon: Group that will have sleeve gastrectomy performed using the Ethicon Echilon powered stapler with absorbable polymer membrane staple line reinforcement. Ethicon Echilon: Surgery performed with Ethicon powered stapler
Period: Overall Study
Arm/Group | Covidien | Ethicon
Started | 30 | 32
Completed | 30 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No information was analyzed for the study and it was closed out in 2019
Groups:
- Total: Total of all reporting groups
Arm/Group | Covidien | Ethicon | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 32 | 62
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 28 | 54
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 15 | 16 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 11 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 32 | 62

OUTCOME MEASURES:

1. Primary Outcome: Time
Description: Time to create sleeve.
Time Frame: Time from first staple firing to last staple firing, for up to 5 hours
Population: Data not collected due to study termination prior to participants' assessment at this time points.
Arm/Group | Covidien | Ethicon
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Staple Firings With Technical Difficulties
Description: Percent of staple firings with technical difficulties
Time Frame: Time from first staple firing to last staple firing, for up to 5 hours
Population: Data not collected due to study termination prior to participants' assessment at this time point.
Arm/Group | Covidien | Ethicon
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Load Time
Description: Time to load staple cartridges
Time Frame: Time from first staple firing to last staple firing, for up to 5 hours
Population: Data not collected due to study termination prior to participants' assessment at this time point.
Arm/Group | Covidien | Ethicon
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Intra-operative Staple Line Bleeding
Description: Will note any incidental bleeding along staple line and how many maneuvers were needed to control it. Measured as: 1) None, 2) Single therapy, 3) Multiple therapy (Any combination of hemostatic modalities)
Time Frame: Time from first staple firing to end of the case, for up to 5 hours
Population: Data not collected due to study termination prior to participants' assessment at this time point.
Arm/Group | Covidien | Ethicon
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Weight Loss
Description: Weight loss in percent excess body weight loss at 3 weeks, 6 weeks, 3 months, 6 months, and up to 1 year
Time Frame: Pre-operative appointment to up to 1 year post-operative, for up to 1 year after sleeve creation
Population: Data not collected due to study termination prior to participants' assessment at this time point.
Arm/Group | Covidien | Ethicon
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Leak Rates
Description: Staple line leak rates
Time Frame: Immediate post-operative period to conclusion of study, for up to 5 hours
Population: Data not collected due to study termination prior to participants' assessment at this time point.
Arm/Group | Covidien | Ethicon
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Readmissions
Description: Hospital readmissions or emergency room visits; Will note reason for readmission
Time Frame: Immediate post-operative period to conclusion of study, for up to 30 days after sleeve creation
Population: Data not collected due to study termination prior to participants' assessment at this time point.
Arm/Group | Covidien | Ethicon
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Sleeve-related Complications Requiring Surgery, Recorded as Yes or no
Description: Will note intervention required and indication; reasons include, but are not limiting to, staple line leak, hematoma, abscess, prolonged tachycardia suspicious for intra-abdominal pathology
Time Frame: Immediate post-operative period to conclusion of study, for up to 1 year after sleeve creation
Population: Data not collected due to study termination prior to participants' assessment at this time point.
Arm/Group | Covidien | Ethicon
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: No Pre-operative EGD (listed in protocol as inclusion criteria). A revised protocol to address this change in inclusion criteria was previously approved under Amendment #3.
Arm/Group | Covidien | Ethicon
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 0/30 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-07-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT02731079/Prot_SAP_001.pdf
  • Informed Consent Form (2016-09-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT02731079/ICF_002.pdf